CLINICAL TRIAL: NCT04799171
Title: Aging and the Mitochondrial Response to Exercise Training, Measured by Noninvasive 31P Magnetic Resonance Spectroscopy (MoTrMito)
Brief Title: Aging and the Mitochondrial Response to Exercise Training, Measured by Noninvasive 31P Magnetic Resonance Spectroscopy
Acronym: MoTrMito
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Colorado, Denver (Other); University of Pittsburgh (Other); The University of Texas Health Science Center at San Antonio (Other); AdventHealth Translational Research Institute (Other); Stanford University (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Owen Carmichael, Director Biomedical Imaging Center, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PBRC 20-03
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-10

CONDITIONS: Physical Activity
Keywords: Isometric contraction exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Young Adults (Age group 18-39) (Active Comparator): 31P-Magnetic Resonance Spectroscopy exam on one thigh to measure mitochondrial capacity non-invasively after exercise training.
  Interventions: Other: Isometric Contraction Exercise - Young Adults (Age group 18-39)
- Middle Aged Adults (Age group 40-59) (Active Comparator): 31P-Magnetic Resonance Spectroscopy exam on one thigh to measure mitochondrial capacity non-invasively after exercise training.
  Interventions: Other: Isometric Contraction Exercise - Middle Age Adults (Age group 40-59)
- Old Adults (Age group >60) (Active Comparator): 31P-Magnetic Resonance Spectroscopy exam on one thigh to measure mitochondrial capacity non-invasively after exercise training.
  Interventions: Other: Isometric Contraction Exercise - Old Adults (Age group >60)

INTERVENTIONS:
Other: Isometric Contraction Exercise - Young Adults (Age group 18-39) — Subjects will be asked to lie supine on MRI table with the 31P surface coil placed over the right vastus lateralis, and straps to immobilize the leg. At the start of the scan session, the investigators will instruct the participant on the isometric contraction exercise and coach the participant through a demonstration. The average flexion repetition time is on the order of 1.5 s for a 30 s duration at maximum kick intensity.
  Arms: Young Adults (Age group 18-39)
Other: Isometric Contraction Exercise - Middle Age Adults (Age group 40-59) — Subjects will be asked to lie supine on MRI table with the 31P surface coil placed over the right vastus lateralis, and straps to immobilize the leg. At the start of the scan session, the investigators will instruct the participant on the isometric contraction exercise and coach the participant through a demonstration. The average flexion repetition time is on the order of 1.5 s for a 30 s duration at maximum kick intensity.
  Arms: Middle Aged Adults (Age group 40-59)
Other: Isometric Contraction Exercise - Old Adults (Age group >60) — Subjects will be asked to lie supine on MRI table with the 31P surface coil placed over the right vastus lateralis, and straps to immobilize the leg. At the start of the scan session, the investigators will instruct the participant on the isometric contraction exercise and coach the participant through a demonstration. The average flexion repetition time is on the order of 1.5 s for a 30 s duration at maximum kick intensity.
  Arms: Old Adults (Age group >60)

SUMMARY:
The goal of the study is to determine whether aerobic or resistant exercise can improve in vivo mitochondrial capacity of skeletal muscle cells similarly in healthy younger, middle aged and older adults. This confers long-term changes in this tissue which in-turn contribute to improved metabolic health and functional capacity through epigenetic regulation of novel exercise response genes.

DETAILED DESCRIPTION:
The goal of the study is to understand the biological pathways and molecules driving the exercise response variation of the muscle mitochondria in vivo to elucidate the underlying mechanisms for the health benefits of exercise training in young, middle aged and older adults. This knowledge will improve investigators understanding of biological basis for targeted "precision medicine" exercise and non-exercise interventions to improve age related conditions. The mitochondrial capacity measurement via non-invasive 31P magnetic resonance spectroscopy (31-MRS) will provide a tangible link between the two primary foci of the parent MoTrPAC study: molecular drivers of exercise response and key phenotypic health outcomes.

ELIGIBILITY:
Inclusion Criteria:

ADULT PARTICIPANT INCLUSION CRITERIA - YOUNG PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrMito Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged 18 - 39 y
* Body Mass Index (BMI) >19 to <35 kg/m2

ADULT PARTICIPANT INCLUSION CRITERIA - MIDDLE AGE PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrMito Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged 40 - 59 y
* Body Mass Index (BMI) >19 to <35 kg/m2

ADULT PARTICIPANT INCLUSION CRITERIA - OLD AGE PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrMito Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged >=60 y
* Body Mass Index (BMI) >19 to <35 kg/m2

Exclusion Criteria:

ADULT PARTICIPANT EXCLUSION CRITERIA

* Exclusion criteria are confirmed by either self-report (i.e., medical and medication histories reviewed by a clinician), screening tests performed by the MoTrMito study team at each clinical site, and/or clinician judgement as specified for each criterion.

Diabetes (self-report and screening tests)

* Treatment with any hypoglycemic agents (self-report) or A1c >6.4 (screening test; may reassess once if 6.5-6.7)
* Fasting glucose >125 (screening test; may reassess once)
* Use of hypoglycemic drugs (e.g., metformin) for non-diabetic reasons (self-report)

Abnormal bleeding or coagulopathy (self-report)

* History of a bleeding disorder or clotting abnormality

Thyroid disease (screening test)

* Thyroid Stimulating Hormone (TSH) value outside of the normal range for the laboratory
* Individuals with hypothyroidism may be referred to their primary care provider (PCP) for evaluation and retested; any medication change must be stable for ≥3 months prior to retesting
* Individuals with hyperthyroidism are excluded, including those with normal TSH on pharmacologic treatment

Pulmonary (self-report)

* Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD)

Metabolic bone disease (self-report)

* History of non-traumatic fracture from a standing height or less
* Current pharmacologic treatment for low bone mass or osteoporosis, other than calcium, vitamin D, or estrogen

Estrogens, progestins (self-report)

* Supplemental, replacement or therapeutic use of estrogens or progestins within the last 6 months, other than birth control or to control menopausal symptoms

Pregnancy (screening test) and pregnancy-related conditions (self-report)

* Pregnant - pregnancy test performed on day of DXA scan in women of child-bearing potential
* Post-partum during the last 12 months
* Lactating during the last 12 months
* Planning to become pregnant during the participation period

Elevated blood pressure readings (screening test)

* Aged <60 years: Resting Systolic Blood Pressure (SBP) ≥140 mmHg or Resting Diastolic Blood Pressure (DBP) ≥90 mmHg
* Aged ≥60 years: Resting SBP ≥150 mmHg or Resting DBP ≥90 mmHg
* Reassessment of BP during screening will be allowed to ensure rested values are obtained

Cardiovascular (self-report, screening test, and clinician judgement)

* Congestive heart failure, coronary artery disease, significant valvular disease, congenital heart disease, serious arrhythmia, stroke, or symptomatic peripheral artery disease (self-report, screening test)
* Specific criteria used to determine whether a volunteer can undergo the screening Cardiopulmonary Exercise Test (CPET) follow the American Heart Association (AHA) Criteria [54]
* Inability to complete the CPET

Abnormal blood lipid profile (screening test)

* Fasting triglycerides >500 mg/dL
* Low-density lipoprotein cholesterol (LDL-C) >190mg/dL

Cancer (self-report)

* History of cancer treatment (other than non-melanoma skin cancer) and not "cancer-free" for at least 2 years
* Anti-hormonal therapy (e.g., for breast or prostate cancer) within the last 6 months

Chronic infection (self-report)

* Infections requiring chronic antibiotic or anti-viral treatment
* Human Immunodeficiency Virus
* Individuals successfully treated for hepatitis C and virologically negative for at least 6 months are not excluded
* Liver enzyme tests (Alanine transaminase, Aspartate transaminase) (screening test) >2 times the laboratory upper limit of normal
* Reassessment during screening may be allowed under some conditions (e.g., recent use of acetaminophen)
* Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting

Chronic renal insufficiency (screening test)

* Estimated glomerular filtration rate <60 mL/min/1.73 m2 from serum creatinine (mg/dL) by the Chronic Kidney Disease Epidemiology Collaboration equation
* Reassessment may be allowed under some conditions (e.g., questionable hydration status or other acute renal insult)

Hematocrit (screening test)

* Hematocrit >3 points outside of the local normal laboratory ranges for women and men Reassessment may be allowed under certain conditions
* Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting
* Individuals with known thalassemia trait may be included (despite having >3 points outside of the local normal laboratory ranges), upon approval from their PCP or a hematologist

Blood donation (self-report)

* Whole blood donation in the last 3 months or plans for blood donation during the entire protocol period
* Platelet or plasma donation in the last week or plans for platelet or plasma donation during the entire protocol period

Autoimmune disorders (self-report)

* Individuals receiving any active treatment (including monoclonal antibodies) within the last 6 months

Alcohol consumption (self-report)

* More than 7 drinks per week for women
* More than 14 drinks per week for men
* History of binge drinking (≥5 drinks for males or ≥4 drinks for females in a 2-hour period more than once per month)

Tobacco (self-report)

* Self-reported use ≥3 days/week of tobacco or e-cigarette/e-nicotine products

Marijuana (self-report)

* Self-reported use ≥3 days/week in any form

Shift workers (self-report)

* Night shift work in the last 6 months
* Planning night shift work during the study period

Cognitive status (screening)

* Unable to give consent to participate in and safely complete the protocol, as based on the judgement of the local investigator

Psychiatric illness (self-report and screening test)

* Hospitalization for any psychiatric condition within one year (self-report)
* Center for Epidemiological Studies-Depression Scale (CESD) score ≥16 [55] (screening test)

Weight change (self-report)

* Weight change (intentional or not) over the last 6 months of >5% of body weight
* Plan to lose or gain weight during the study
* Lidocaine or other local anesthetic (self-report)
* Known allergy to lidocaine or other local anesthetic

Other (clinician judgement)

* Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric or other conditions that, in the opinion of the local clinician, would preclude participation and successful completion of the protocol
* Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol

EXCLUSIONS FOR MEDICATION USE

* Use of any new drug in the last 3 months
* Dose change for any drug in the last within 3 months

Cardiovascular

* Beta blockers and centrally acting anti-hypertensive drugs (clonidine, guanfacine and alpha-methyl-dopa)

Anticoagulants (coumadin or Direct Oral Anticoagulants)

Antiarrhythmic drugs: amiodarone, dronaderone, profafenone, disopyrimide, quinidine

Antiplatelet drugs (other than aspirin ≥100 mg/day): dipyridamole, clopidogrel, ticagrelor

Lipid-lowering medications

* Participants who volunteer to stop lipid-lowering medications for the duration of the study are allowed; inclusion requires lipid-lowering medication to be stopped for 3 months and participant re-evaluated for LDL-C eligibility

Psychiatric drugs

* Chronic use of medium or long-acting sedatives and hypnotics (short-acting non-benzodiazepine sedative-hypnotics are allowed)
* All benzodiazepines
* Tricyclic antidepressants at a dose ≥75 mg total dose per day
* Two or more drugs for depression
* Mood stabilizers

Antiepileptic drugs

* Stimulants, Attention-Deficit/Hyperactivity Disorder (ADHD) drugs

Muscle relaxants

* Methacarbamol; cyclobenzaprine; tizanidine; baclofen

Pulmonary, inflammation

Chronic oral steroids

* Burst/taper oral steroids more than once in the last 12 months
* B2-agonists allowed if on stable dose at least 3 months

Genitourinary

* Finasteride or dutasteride
* Daily phosphodiesterase type 5 inhibitor use

Hormonal

* Testosterone, dehydroepiandrosterone, anabolic steroids
* Anti-estrogens, anti-androgens
* Growth hormone, insulin like growth factor-I, growth hormone releasing hormone
* Any drugs used to treat diabetes mellitus or to lower blood glucose
* Metformin for any indication
* Any drugs used specifically to induce weight loss
* Any drugs used specifically to induce muscle growth/hypertrophy or augment exercise-induced muscle hypertrophy
* Pain/inflammation

Narcotics and narcotic receptor agonists

* Regular use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen ≥3 days per week
* Other

Anti-malarials

* Low-potency topical steroids if ≥10% of surface area using rule of 9s
* Any other medications that, in the opinion of local clinicians, would negatively impact or mitigate full participation and completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Pre-training 31P MRS measurement - Phosphocreatine recovery rate | Baseline visit - before any muscle biopsies or exercise training.
  The plot of PCr peak height vs. time will be fitted with a mono-exponential equation whose free parameters are the recovery time constant (tau) and scaling coefficients. Percent change in tau between pre- and post-intervention scans will be our primary measurement of the maximal mitochondrial capacity response to exercise training.
Post-training 31P MRS measurement - Phosphocreatine recovery rate | After week 12 visit - after all muscle biopsies and exercise training.
  The plot of PCr peak height vs. time will be fitted with a mono-exponential equation whose free parameters are the recovery time constant (tau) and scaling coefficients. Percent change in tau between pre- and post-intervention scans will be our primary measurement of the maximal mitochondrial capacity response to exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Owen T Carmichael, PhD, Principal Investigator — Director, Biomedical Imaging Center, PBRC
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
As a MoTrPAC ancillary study, we will comply with all regulations of the MoTrPAC Ancillary Study Committee regarding sharing of data generated from MoTrPAC participants. We will follow up on any data irregularities identified by the Bioinformatics Core as part of their data cleaning process. The Bioinformatics Core will then make our MRS summary data ancillary study data to the community together with the MoTrPAC main study data and data from any other ancillary studies that arise. We are familiar with the NIH policies regarding data sharing, and during our data transfer to the main MoTrPAC study we will comply with local, state, and federal laws, such as the Privacy Rule, a Federal regulation under the Health Insurance Portability and Accountability Act (HIPAA).